CLINICAL TRIAL: NCT01385098
Title: Preoperative Vitamin D Status and Efficacy of Therapeutic Vitamin D Supplementation Postoperatively in Bariatric Surgery Patients
Brief Title: Efficacy of Vitamin D Supplementation in Bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vadim Sherman, MD (Other)
Collaborators: Texas Woman's University (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Vadim Sherman, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005625; 0311-0034 (Other: HMRI IRB)
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Obesity; Vitamin D Deficiency
Keywords: Vitamin D; Bariatric surgery; Roux-en Y surgery; Gastric sleeve surgery; Parathyroid Hormone
MeSH Terms: conditions — Obesity; Vitamin D Deficiency | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D3 and Calcium (Experimental): Dietary supplement of vitamin D3 and calcium
  Interventions: Dietary Supplement: Vitamin D3 and Calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D3 and Calcium — 1500 mg of calcium citrate plus 1000 IU of vitamin D3 and 1000 IU of vitamin D3 bariatric supplements per day
  Other Names: Celebrate ® calcium citrate plus vitamin D3; Celbrate ® multi-vitamin

SUMMARY:
As the use of bariatric surgery for treatment of extreme obesity adults continues to rise, clinicians must be aware of pre-existing nutritional deficiencies in overweight and obese patients. Nutritional deficiencies are common in patients undergoing bariatric surgery and these deficiencies should be detected and addressed early to avoid post-operative complications. To improve long-term outcomes following bariatric surgery, nutritional screening and prescribing appropriate supplementation to prevent nutrient deficiencies is needed. Vitamin D deficiency is common following bariatric surgery and has been reported to occur in 50-80% bariatric patients.The goal of this pilot study is to help develop nutrient supplementation interventions following two types of bariatric surgery: Roux-en Y gastric bypass and sleeve gastrectomy.

Recently, several studies in adults have revealed an inverse relationship between body fat and blood 25-hydroxyvitamin D3 [25(OH)D] levels, the relevant marker of low vitamin D status. Although vitamin D is well known for its essential role in bone metabolism and calcium homeostasis, increasing evidence is linking vitamin D to obesity. This study will evaluate vitamin D status during post operative daily supplementation of 2,000 IU of vitamin D3 and 1500 mg of calcium through assessment of changes in serum 25(OH)D, parathyroid hormone (PTH), calcium and phosphorus at baseline, 4 weeks, and 12 weeks following surgery. The dietary contribution of vitamin D and calcium will be estimated by food records analyzed using the University of Minnesota 2010 Nutrition Data System for Research (NDSR) program.

Primary Hypothesis: Daily supplementation with 2,000 IU of vitamin D3 for 12 weeks will significantly increase mean serum 25(OH)D levels in obese subjects following bariatric surgery compared to baseline levels.

Secondary Hypothesis: The percent response above baseline to daily supplementation with 2,000 IU of vitamin D3 will significantly differ between Roux-en Y and sleeve gastrectomy patients.

DETAILED DESCRIPTION:
The prospective pilot study is designed to evaluate vitamin D status pre-operatively and post-operatively in 37 female patients undergoing either Roux-en Y gastric bypass or sleeve gastrectomy at The Methodist Hospital with 32 patients expecting to complete the 12 week trial. Women scheduled for either of these two types of bariatric surgery will be considered for inclusion in the pilot study. Based on previous research experience at The Methodist Hospital, the majority of bariatric patients are women. No children are treated at the Methodist Hospital bariatric center.

Subjects will be excluded if they have evidence of vitamin D deficiency (25(OH)D <20 ng/mL), hypercalcemia (calcium > 2.63 mmol/L), hypocalcemia (calcium < 1.75 mmol/L), renal insufficiency (GFR < 50 ml/min), or a history of primary hyperparathyroidism or renal tubular acidosis. Participants will be excluded if they take medications that interfere with vitamin D metabolism, have significant sun exposure, plan to travel to sunny climates during the study, or a history of hypercalcemia.

Baseline measures of serum 25(OH)D, PTH, calcium and phosphorus will be obtained. Values will be determined one week prior to surgery and during the follow-up visit at 12 weeks postoperatively. In addition, 25(OH)D will be measured at the 4th week post-operative clinic visit. Baseline information obtained will include age, height (centimeter), weight (kilogram), body mass index, sex, and race or ethnicity. A full medication list and medical history to identify any co-morbid conditions will be collected. Participants will be instructed to avoid traveling to sunny locations during the 12 week study.

Laboratory measurements pre-operative: 25(OH)D, PTH, CBC/Diff, glucose, calcium, albumin, total protein, sodium, potassium, CO2, BUN, creatinine, ALP, ALT, AST, bilirubin, lipid panel, ferritin, folate, iron, total iron binding capacity, hemoglobin A1c, insulin, vitamin B12, PT/PTT, TSH, HCG, C-reactive protein.

Laboratory measurements at week 4: 25(OH)D

Laboratory measurements at week 12: 25(OH)D, PTH, CBC/Diff, glucose, calcium, albumin, total protein, sodium, potassium, CO2, BUN, creatinine, ALP, ALT, AST, bilirubin, lipid panel, ferritin, folate, total iron binding capacity, vitamin B12, and TSH.

Nutrient intake assessments: Dietary intake of macronutrients, vitamin D, calcium, and other micronutrients will be assessed using the University of Minnesota 2010 Nutrition Data System for Research (NDSR) program. NDSR is a comprehensive nutrient calculation software program used for research purposes. The NDSR database contains values for 160 nutrients and includes more than 18,000 foods.

Participants' baseline laboratory will be used to measure the response to vitamin D and calcium supplementation over the course of 12 weeks. Bariatric patients participating in the study will be instructed to take a total of 1500 mg of calcium (as calcium citrate) plus 1000 IU of vitamin D3 as three chewable tablets (Celebrate ®). An addition 1000 IU of vitamin D3 per day will be taken as two chewable multi-vitamin bariatric supplements (Celebrate ®). Supplement compliance will be assessed by daily written records and inspection of supplement bottle containers at each clinic visit.

Serum 25(OH)D will be measured by ARUP Laboratories (Salt Lake City, UT, USA) using a chemiluminescent immunoassay. Serum calcium and phosphorus will be determined by The Methodist Hospital Clinical Chemistry Department as part of the standard bariatric protocol comprehensive metabolic panel. Intact PTH (iPTH) assays will be performed using the ADVIA Centaur ® XP Immunoassay System.

Vitamin D deficiency will be defined as 25(OH)D levels less than 20 ng/mL (50 nmol/L) and vitamin D insufficiency as 21 to 29 ng/mL (50 to 80 nmol/L). Secondary hyperparathyroidism will be defined as iPTH ≥ 70 ng/L. An increase in serum intact PTH level will be taken to be indicative of a possible negative calcium balance or a vitamin D deficiency (or both). Hypercalcemia will be defined as calcium > 2.63 mmol/L.

Statistical analysis:

Primary Hypothesis: Daily supplementation with 2,000 IU of vitamin D3 for 12 weeks will significantly increase mean serum 25(OH)D levels in obese subjects following bariatric surgery compared to baseline levels.

Secondary Hypothesis: The percent response above baseline to daily supplementation with 2,000 IU of vitamin D3 will significantly differ between Roux-en Y and sleeve gastrectomy patients.

Subject Withdrawal:

Participants will be withdrawn from the study if serum 25(OH)D levels are identified as within the deficient range so that the patient can receive needed treatment. A vitamin D deficiency will be defined as 25(OH)D concentrations less than 20 ng/mL (50 nmol/L) and vitamin D insufficiency as 21 to 29 ng/mL. In addition, if an abnormally high level of 25(OH)D is obtained (200 ng/mL or 500 nmol/L), we will have the 25(OH)D measurement repeated. If the second test is confirmed to be high, then we will withdraw that particular patient from the study for medical follow-up. If we find a trend of excess vitamin D among participants, however, we will re-evaluate and consider termination of the study.

ELIGIBILITY:
Inclusion Criteria: Adult female obese patients undergoing either Roux-en Y gastric bypass or sleeve gastrectomy at The Methodist Hospital may participate in the study. Obese patients with a body mass index (BMI) > 40 or BMI >35 with a co-morbidity will be eligible.

-

Exclusion Criteria:Subjects will be excluded if they have evidence of vitamin D deficiency (< 20 ng/mL), hypercalcemia (calcium > 2.63 mmol/L), hypocalcemia (calcium < 1.75 mmol/L), renal insufficiency (GFR < 50 ml/min), or a history of primary hyperparathyroidism or renal tubular acidosis.Participants will be excluded if they take medications that interfere with vitamin D metabolism, have significant sun exposure, plan to travel to sunny climates during the study, or a history of hypercalcemia.

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Miller, MD, Study Chair — The Methodist Hospital Research Institute; Vadim Sherman, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlin AM, Rao DS, Yager KM, Parikh NJ, Kapke A. Treatment of vitamin D depletion after Roux-en-Y gastric bypass: a randomized prospective clinical trial. Surg Obes Relat Dis. 2009 Jul-Aug;5(4):444-9. doi: 10.1016/j.soard.2008.08.004. Epub 2008 Aug 14. PMID 18996761
- [Background] Compher CW, Badellino KO, Boullata JI. Vitamin D and the bariatric surgical patient: a review. Obes Surg. 2008 Feb;18(2):220-4. doi: 10.1007/s11695-007-9289-6. Epub 2008 Jan 5. PMID 18176832
- [Background] Gemmel K, Santry HP, Prachand VN, Alverdy JC. Vitamin D deficiency in preoperative bariatric surgery patients. Surg Obes Relat Dis. 2009 Jan-Feb;5(1):54-9. doi: 10.1016/j.soard.2008.07.008. Epub 2008 Jul 24. PMID 18848507
- [Background] Mechanick JI, Kushner RF, Sugerman HJ, Gonzalez-Campoy JM, Collazo-Clavell ML, Guven S, Spitz AF, Apovian CM, Livingston EH, Brolin R, Sarwer DB, Anderson WA, Dixon J. American Association of Clinical Endocrinologists, The Obesity Society, and American Society for Metabolic & Bariatric Surgery Medical Guidelines for Clinical Practice for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient. Surg Obes Relat Dis. 2008 Sep-Oct;4(5 Suppl):S109-84. doi: 10.1016/j.soard.2008.08.009. Epub 2008 Aug 19. PMID 18848315
- [Background] Gastrointestinal surgery for severe obesity: National Institutes of Health Consensus Development Conference Statement. Am J Clin Nutr. 1992 Feb;55(2 Suppl):615S-619S. doi: 10.1093/ajcn/55.2.615s. PMID 1733140
- [Result] Moore CE, Sherman V. Vitamin D supplementation efficacy: sleeve gastrectomy versus gastric bypass surgery. Obes Surg. 2014 Dec;24(12):2055-60. doi: 10.1007/s11695-014-1261-7. PMID 24748475
- [Derived] Chakhtoura MT, Nakhoul NF, Akl EA, Safadi BY, Mantzoros CS, Metzendorf MI, El-Hajj Fuleihan G. Oral vitamin D supplementation for adults with obesity undergoing bariatric surgery. Cochrane Database Syst Rev. 2024 Oct 1;10(10):CD011800. doi: 10.1002/14651858.CD011800.pub2. PMID 39351881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D3 and Calcium
Started | 37
Completed | 23 (14 subjects did not complete. 4 subjects loss to follow-up & 10 subjects could not tolerate suppl.)
Not Completed | 14
Not completed — Adverse Event | 10
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Number of completers
Arm/Group | Vitamin D3 and Calcium
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
BMI, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 46.3 (8.1)
Body weight, lb [Mean (Standard Deviation); unit: lb] | 278 (52)
Excess body weight, lb [Mean (Standard Deviation); unit: lb] | 128 (47)
Surgery type [Count of Participants; unit: Participants]
  Sleeve Gastrectomy | 11
  Roux-Y Gastric Bypass | 12

OUTCOME MEASURES:

1. Primary Outcome: Vitamin D Concentrations, Pre Operative and Post Bariatric Surgery Following 12 Weeks of Vitamin D Supplementation
Description: Serum 25(OH)D ng/ml levels at baseline and 12 weeks following bariatric surgery
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D3 and Calcium
Number analyzed (Participants) | 23
ng/mL
  Preoperative | 19.1 (9.0)
  12 weeks | 27.2 (8.4)
Statistical Analysis 1: Comparison: Vitamin D3 and Calcium; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Serum 25-hydroxyvitamin D Levels at Baseline and 12 Weeks of Daily Vit D Supplementation Post Roux-en Y OR Sleeve Gastrectomy
Description: We anticipate that vitamin D supplementation of Roux-en Y bariatric surgery patients will be less effective in improving or maintaining vitamin D status.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Sleeve Gastrectomy; Roux-Y Gastric Bypass: Dietary supplement of vitamin D3 and calcium
  Vitamin D3 and Calcium: 1500 mg of calcium citrate plus 1000 IU of vitamin D3 and 1000 IU of vitamin D3 bariatric supplements per day
Arm/Group | Sleeve Gastrectomy | Roux-Y Gastric Bypass
Number analyzed (Participants) | 11 | 12
ng/mL
  Preoperative | 18.5 (9.6) | 19.6 (8.3)
  12 Weeks | 26.3 (9.6) | 28.1 (7.6)
Statistical Analysis 1: Comparison: Sleeve Gastrectomy; Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney) — Change from preoperative to 12 weeks
Statistical Analysis 2: Comparison: Roux-Y Gastric Bypass; Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney) — Change from preoperative to 12 weeks

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Vitamin D3 and Calcium
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No